CLINICAL TRIAL: NCT02781090
Title: RCT of an Internet Cessation Program Plus Online Social Network for HIV+ Smokers
Acronym: PSFW+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Westat (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-4723
Record Dates: First submitted 2016-04-28; First posted 2016-05-24 (Estimated); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Tobacco Use Disorder; HIV
Keywords: HIV; Tobacco; Cigarette; Smoking; Social Network; Internet; Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Positively Smoke Free on the Web (PSFW+) (Experimental): Participants were assigned to the multimodal PSFW+ interactive web-based behavioral intervention hosted within an online social network.
  PSFW+: PSFW+ is an intensive eight session motivational/educational web-program, based on social cognitive theory, designed to promote cessation among HIV-infected smokers. It included a professionally administered social network/online support community.
  Nicotine polacrilex: All participants were offered a 3-month supply of nicotine patches
  Interventions: Behavioral: PSFW+; Drug: Nicotine polacrilex
- American Heart Association Getting Healthy (AHA) (Placebo Comparator): Participants were assigned to the AHA Getting Healthy web-based control intervention program (the AHA later changed in name from "Getting Healthy" to "My Life's Check, Life's Simple 7"
  AHA: The AHA Getting Healthy website is an attention-matched, health-promoting, seven-module website developed by the American Heart Association to encourage healthy behaviors in the general population
  Nicotine polacrilex: All participants were offered a 3-month supply of nicotine patches
  Interventions: Behavioral: AHA; Drug: Nicotine polacrilex

INTERVENTIONS:
Behavioral: PSFW+ — PSFW+ is an eight session motivational/educational web-program promoting cessation for HIV-infected smokers. It includes a professionally administered social network/online support community.
  Other Names: AHA
  Arms: Positively Smoke Free on the Web (PSFW+)
Behavioral: AHA — The AHA Getting Healthy website is a health-promoting, seven-module website developed by the American Heart Association to encourage healthy behaviors in the general population
  Arms: American Heart Association Getting Healthy (AHA)
Drug: Nicotine polacrilex — All participants, in both study arms, will be offered a 3-month supply of nicotine patches
  Other Names: Nicotine patch

SUMMARY:
This trial will compare the efficacy of Positively Smoke Free on the Web+ (a smoking cessation program + social network for HIV-infected smokers) to the American Heart Association Getting Healthy website in promoting abstinence in a group of HIV-infected smokers. All participants will be offered a three-month supply of nicotine patches.

DETAILED DESCRIPTION:
There are 1.1 million persons living with HIV (PLWH) in the US: 60% smoke cigarettes and 75% are interested in quitting. Two-thirds of PLWH use the Internet, making this a promising avenue to deliver smoking cessation treatment. Almost none are currently accessing smoking cessation interventions designed to meet their specific needs and concerns. Cigarette smoking is responsible for 24%--61% of deaths among PLWH, and 30% of non-AIDS defining malignancies. It is driving the alarming rise in lung cancers in this highly vulnerable population. The lack of access to proven, effective, culturally appropriate tobacco cessation services represents a health disparity of the first order.

Cessation websites offer smokers convenience, low (or no) cost, and anonymity; however, there are no publicly available web-based cessation programs specifically designed for PLWH smokers. Smokers living with HIV have high rates of nicotine dependence, anxiety, depression, loneliness, and substance use. The investigators developed Positively Smoke Free on the Web (PSFW), a theory-driven, culturally tailored web-based program designed to address the specific needs of PLWH smokers. The investigators' NCI-funded R21 pilot of PSFW demonstrated moderate-high levels of adherence and yielded higher 3-month abstinence rates compared to standard care (10% vs. 4%). The investigators' prior research on web-based cessation interventions has shown that smokers who participate in an online community - whether passively reading posts by others or actively engaging in online discussions - are more than twice as likely to achieve abstinence even after controlling for a broad range of covariates. In preparation for the proposed study, the investigators' partners at Truth Initiative (formerly known as the American Legacy Foundation) have enhanced and modernized PSFW by integrating an online community platform (now "PSFW+"), developing a training protocol for PLWH smoker seed users (to provide a critical mass of social network participants), and recruiting and training 11 PLWH smokers for this role. The prototype PSFW+ application has been successfully alpha- and beta-tested in anticipation of the randomized controlled trial.

The investigators propose a study that will compare the efficacy of the PSFW+ smoking cessation website to an attention-matched website promoting cardiovascular health in a randomized controlled trial with repeated measures at baseline, 1, 3, and 6 months. Participants will be N=550 PLWH smokers interested in quitting in the next 30 days. All participants will be offered nicotine replacement therapy. It is hypothesized that PSFW+ will outperform the control condition on the primary outcome of 7-day point prevalence abstinence at 6 months post-randomization. Secondary aims and exploratory analyses will examine theory-driven hypotheses about the mediators and moderators of treatment outcome (e.g., depression, anxiety, social support, loneliness, self-efficacy). Establishing the effectiveness of a web-based smoking cessation program for PLWH that has broad reach and could be scaled to reach PLWH smokers throughout the US would not only represent an enormous advance in the fight against tobacco use in PLWH, but would also provide a clearer understanding of the role of targeted, web-based health interventions in comprehensive HIV care.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 or older
2. current smoking as defined by a validated tobacco use measure
3. laboratory confirmed HIV-infection; 3) residence in commuting distance to the Bronx, NY or Baltimore, MD
4. English language fluency
5. motivation to quit within the next 30 days
6. at least weekly Internet and email access
7. REALM literacy score of 19/66 or above, indicating reading level of at least 4-6 grade (PSFW content was written for this literacy level)
8. willingness to provide informed consent and undergo randomization.

Exclusion Criteria:

1. previous participation in any trial of Positively Smoke Free interventions or use of PSFW+
2. pregnancy
3. contraindication to nicotine replacement therapy
4. current participation in an active smoking cessation treatment (e.g., group therapy, use of pharmacotherapy)
5. PSFW+ seed users will be excluded
6. To avoid study condition contamination and to maintain the statistical independence of subject outcomes, otherwise eligible individuals who are spouses, partners, and/or roommates of study participants will be excluded.

All ineligible patients will receive a Positively Smoke Free smoking cessation brochure and will be encouraged to access nationally-available (free) quitline counseling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shuter, MD, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Johns Hopkins, Baltimore, Maryland
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD at this time.

REFERENCES:
- [Background] Shuter J, Morales DA, Considine-Dunn SE, An LC, Stanton CA. Feasibility and preliminary efficacy of a web-based smoking cessation intervention for HIV-infected smokers: a randomized controlled trial. J Acquir Immune Defic Syndr. 2014 Sep 1;67(1):59-66. doi: 10.1097/QAI.0000000000000226. PMID 25118794
- [Derived] Mdege ND, Shah S, Dogar O, Pool ER, Weatherburn P, Siddiqi K, Zyambo C, Livingstone-Banks J. Interventions for tobacco use cessation in people living with HIV. Cochrane Database Syst Rev. 2024 Aug 5;8(8):CD011120. doi: 10.1002/14651858.CD011120.pub3. PMID 39101506
- [Derived] Shuter J, Chander G, Graham AL, Kim RS, Stanton CA. Randomized Trial of a Web-Based Tobacco Treatment and Online Community Support for People With HIV Attempting to Quit Smoking Cigarettes. J Acquir Immune Defic Syndr. 2022 Jun 1;90(2):223-231. doi: 10.1097/QAI.0000000000002936. PMID 35175971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through provider referrals from the two clinical trial sites, Montefiore Medical Center's Center for Positive Living in the Bronx, NY and Johns Hopkins Bartlett Clinic for Infectious Diseases in Baltimore, MD, between July 2016 and March 2020. Participants were also recruited by direct contact in the clinical waiting areas, and by self-referral in response to study advertisements.
Pre-assignment Details: Of 512 enrolled participants, 506 met inclusion criteria and were randomized into one of the two study arms/groups. Six of the 512 trial enrollees were excluded from the final trial data set for the following reasons: two participants disenrolled immediately following randomization, two participants were ineligible due to seed user status, and two participants were excluded for enrolling in the trial a second time.
Period: 3-Month Follow-Up
Arm/Group | Positively Smoke Free on the Web (PSFW+) | American Heart Association Getting Healthy (AHA)
Started | 255 | 251
Completed | 190 | 194
Not Completed | 65 | 57
Not completed — Missed Visit | 20 | 20
Not completed — Lost to Follow-up | 40 | 34
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Death | 1 | 0
Period: 6-Month Follow-Up
Arm/Group | Positively Smoke Free on the Web (PSFW+) | American Heart Association Getting Healthy (AHA)
Started | 190 | 194
Completed | 169 | 169
Not Completed | 21 | 25
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 20 | 22
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positively Smoke Free on the Web (PSFW+) | American Heart Association Getting Healthy (AHA) | Total
Number analyzed (Participants) | 255 | 251 | 506
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.47 (10.20) | 49.95 (10.63) | 50.21 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 110 | 216
  Male | 149 | 141 | 290
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 46 | 97
  Not Hispanic or Latino | 204 | 205 | 409
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 8 | 10
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 3 | 9 | 12
  Black or African American | 213 | 205 | 418
  White | 36 | 29 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 255 | 251 | 506

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving 7-day Point Prevalence Abstinence From Tobacco Use
Description: The number of participants achieving 7-day Point Prevalence Abstinence (PPA) from tobacco use at 6 months was determined for each study arm. 7-day PPA parameters for this study were based on the number of participants demonstrating biochemically confirmed exhaled carbon monoxide (< 10ppm).
Time Frame: 6 months
Population: Intention to treat (ITT) analysis. Lost to follow-up participants were assumed to be non-abstinent
Measure: Count of Participants; unit: Participants
Arm/Group | Positively Smoke Free on the Web (PSFW+) | American Heart Association Getting Healthy (AHA)
Number analyzed (Participants) | 255 | 251
Participants
  Abstinent | 38 | 22
  Non-Abstinent | 217 | 229

2. Secondary Outcome: Website Satisfaction
Description: Questionnaires were administered to all study participants at 6 months to assess participant satisfaction with the PSFW+ and AHA 'Getting Healthy' website and online tools. Participants were asked to provide feedback regarding their level of satisfaction with the online platform using the following response options: Not at all Satisfied, A little Satisfied, Moderately Satisfied, Very Satisfied, or Extremely Satisfied. Participants responses were aggregated and tabulated.
Time Frame: Up to 6 months
Population: The Overall Number of Participants analyzed for this outcome measure is indicative of satisfaction survey questionnaires completed and received at both the 3 month and the 6 month follow-up visits. Some participants who did not show up for the 3-month visit were successfully recalled for the 6-month visit.
Measure: Number; unit: participants
Groups:
- Positively Smoke Free on the Web (PSFW+): Participants were assigned to the multimodal PSFW+ interactive web-based behavioral intervention hosted within an online social network.
  PSFW+: PSFW+ is an intensive eight session motivational/educational web-program, based on social cognitive theory, designed to promote cessation among HIV-infected smokers. It included a professionally administered social network/online support community.
  Nicotine polacrilex: All participants were offered a 3-month supply of nicotine patches
  PSFW+: PSFW+ is an eight session motivational/educational web-program promoting cessation for HIV-infected smokers. It includes a professionally administered social network/online support community.
  Nicotine polacrilex: All participants, in both study arms, will be offered a 3-month supply of nicotine patches
- American Heart Association Getting Healthy (AHA): Participants were assigned to the AHA Getting Healthy web-based control intervention program (the AHA later changed in name from "Getting Healthy" to "My Life's Check, Life's Simple 7"
  AHA: The AHA Getting Healthy website is an attention-matched, health-promoting, seven-module website developed by the American Heart Association to encourage healthy behaviors in the general population
  Nicotine polacrilex: All participants were offered a 3-month supply of nicotine patches
  AHA: The AHA Getting Healthy website is a health-promoting, seven-module website developed by the American Heart Association to encourage healthy behaviors in the general population
  Nicotine polacrilex: All participants, in both study arms, will be offered a 3-month supply of nicotine patches
Arm/Group | Positively Smoke Free on the Web (PSFW+) | American Heart Association Getting Healthy (AHA)
Number analyzed (Participants) | 206 | 204
participants
  Not at all satisfied | 16 | 16
  A little satisfied | 34 | 45
  Moderately satisfied | 62 | 50
  Very satisfied | 68 | 63
  Extremely satisfied | 25 | 24
  Refused or missing | 1 | 6

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Positively Smoke Free on the Web (PSFW+) | American Heart Association Getting Healthy (AHA)
All-Cause Mortality (participants affected / at risk) | 1/255 | 1/251
Serious Adverse Events (participants affected / at risk) | 0/255 | 0/251
Other Adverse Events (participants affected / at risk) | 0/255 | 0/251

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT02781090/Prot_SAP_000.pdf